CLINICAL TRIAL: NCT00830362
Title: Treatment Implications of Beta-blockade Effects on Memory for Cocaine Craving
Brief Title: Beta-blockade Effects on Memory for Cocaine Craving
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 18285; R21DA025155 (NIH); R21DA025155-01 (NIH); DPMC (Other: NIDA)
Record Dates: First submitted 2009-01-26; First posted 2009-01-27 (Estimated); Results first posted 2012-11-30 (Estimated); Last update posted 2012-11-30 (Estimated); Status verified 2012-09

CONDITIONS: Cocaine Dependence
Keywords: cocaine; cocaine-dependent; propranolol; craving; beta-blockade; cue exposure; drug; addiction; memory; addictive behavior
MeSH Terms: conditions — Cocaine-Related Disorders; Behavior, Addictive | interventions — Propranolol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Propranolol 40mg (Active Comparator)
  Interventions: Drug: Propranolol
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Propranolol — 40 mg administered once
  Arms: Propranolol 40mg
Drug: Placebo — administered once
  Arms: Placebo

SUMMARY:
The purpose of this study is to examine the effects of propranolol versus placebo on responses to cocaine cues in cocaine dependent individuals.

DETAILED DESCRIPTION:
This study will employ cocaine-dependent individuals to investigate the acute effects of propranolol vs. placebo, administered immediately after a retrieval session of cocaine cue exposure, on the subjective and physiological responses occurring during a subsequent test session of cocaine cue exposure. Participants (N=52) will be randomly assigned to receive 40 mg propranolol or placebo immediately after the first of two cocaine cue exposure sessions scheduled to occur on consecutive days of an inpatient stay at MUSC's General Clinical Research Center (GCRC). The first session will serve as a retrieval session where cocaine cue exposure will putatively elicit retrieval and reconsolidation of memories about the association between the cues and cocaine administration; the second session of cocaine cue exposure will be a test session to examine the potential modulatory role of propranolol on the reconsolidated memories putatively elicited during the previous cue exposure session. It is assumed that changes in craving and physiological reactivity during the test session will reflect propranolol's effects on memory reconsolidation processes elicited by cue exposure during the retrieval session. Medications will be administered in a double-blind fashion. Craving and physiological arousal (heart rate, skin conductance, blood pressure) will be obtained at baseline and at regular intervals during and after both cue exposure sessions. Approximately 7 days following discharge from the inpatient stay at the GCRC, participants will return to the GCRC to undergo a 1-week follow-up cue exposure session that will be identical to the previous two sessions (no medications will be administered). The goal of the follow-up will be to examine if any craving and/or physiological reactivity differences identified during the test session were sustained and to assess if the groups differed in their cocaine use during the intervening 7-day period.

ELIGIBILITY:
Inclusion Criteria:

* Current cocaine dependence (within past month)
* Able to provide informed consent
* Use of birth control by female participants (barrier methods, surgical sterilization, IUD, or abstinence)
* Live within 50-mile radius of research site
* Consent to remain abstinent from all drugs of abuse (except nicotine) for 24 hours prior to inpatient admission and follow-up assessment
* Consent to random assignment to propranolol or placebo

Exclusion Criteria:

* Women who are pregnant, nursing or are of childbearing potential and not practicing/using birth control
* Evidence or history of significant hematological, endocrine, cardiovascular, pulmonary, renal, gastrointestinal or neurological disease
* Significant liver impairment
* History of or current psychotic disorder, current severe major depressive disorder, bipolar affective disorder or a severe anxiety disorder
* Currently taking anti-arrhythmic agents, psychostimulants or other agents known to interfere with heart rate and skin conductance monitoring
* Known or suspected hypersensitivity to propranolol
* Individuals taking medications that could adversely interact with the study medication, including, but not limited to albuterol, insulin, or significant inhibitors of CYP2D6
* Individuals with bronchial asthma or chronic obstructive pulmonary disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2009-02; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Saladin, Ph.D., Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Individuals who met DSM-IV criteria for current cocaine dependence (within the past month) but who were not dependent on any other substance, with the exception of nicotine, served as participants. The primary method of recruitment was media advertisement (radio, local papers) which ran from January of 2009 until July of 2011.
Pre-assignment Details: Exclusion criteria included severe psychiatric comorbidity (e.g., psychotic disorder, bipolar disorder, severe major depressive disorder with suicidal ideation) or medical illness or use of medications that might interact with propranolol. Individuals with other substance dependence (with exception of nicotine) were also excluded at initial visit.
Groups:
- Propranolol 40mg: Propranolol : 40 mg administered once. The subjects whose data we analyzed upon study completion who received propranolol were those that received the medication and completed BOTH the test and retrieval sessions (Session 1 and 2). Our N=50 that we report in the protocol section the total number of participants (from both the propranolol and placebo groups) that were analyzed.
- Placebo: Placebo : administered once. The subjects whose data we analyzed upon study completion who received placebo were those that received the medication and completed BOTH the test and retrieval sessions (Session 1 and 2). Our N=50 that we report in the protocol section the total number of participants (from both the propranolol and placebo groups) that were analyzed.
Period: Overall Study
Arm/Group | Propranolol 40mg | Placebo
Started | 27 (They received Propranolol and completed Test Session (Session 1). One subject left after day 1.) | 24 (They received Propranolol and completed Test Session (Session 1). One subject left after day 1.)
Completed Sessions 1 and 2 | 26 (Received propranolol and completed both Test and Retrieval sessions (Session 1 and 2).) | 24 (Received palcebo and completed both Test and Retrieval sessions (Session 1 and 2).)
Completed | 23 (The enrolled subjects that completed all 3 testing sessions (were not lost to follow-up).) | 20 (The enrolled subjects that completed all 3 testing sessions (were not lost to follow-up).)
Not Completed | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Propranolol 40mg: Propranolol : 40 mg administered once. The subjects analyzed who received propranolol were those that received the medication and completed both the test and retrieval sessions (Test Day 1 and 2).
- Placebo: Placebo : administered once. The subjects analyzed who received placebo were those that received the sugar pill and completed both the test and retrieval sessions (Test Day 1 and 2).
- Total: Total of all reporting groups
Arm/Group | Propranolol 40mg | Placebo | Total
Number analyzed (Participants) | 26 | 24 | 50
Age Continuous [Mean (Standard Deviation); unit: years] | 39.1 (1.6) | 40.8 (2.0) | 39.9 (1.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 8 | 17
  Male | 17 | 16 | 33

OUTCOME MEASURES:

1. Primary Outcome: Single Item Craving Test Session Difference Scores
Description: Mean of the difference of Session 1 and Session 2 cocaine craving scores (Session 2-Session 1). Found by using our Single Item Craving (SIC) scale. A study team member asks the participant to verbally report the level of craving they were experiencing using values between 0 and 100, with 0 representing no craving and 100 extreme craving. The difference score was found by subtracting session 1 mean SICs during cue exposure from session 2 mean SICs during cue exposure. Therefore the mean of the difference could have ranged anywhere from -100 to 100. Negative mean difference scores reflect a decrease in craving for cocaine from session 1 (test) to session 2 (retrieval). The lower the mean difference score, the greater the decrease in craving.
Time Frame: Both days of cue exposure
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Propranolol 40mg | Placebo
Number analyzed (Participants) | 26 | 24
units on a scale | -25.0 (4.5) | -10.5 (4.7)

ADVERSE EVENTS:
Arm/Group | Propranolol 40mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/24
Other Adverse Events (participants affected / at risk) | 0/27 | 0/24

LIMITATIONS AND CAVEATS:
Lack of a "no retrieval" control group. Lack of determination of plasma propranolol levels following the medicated retrieval session. The sample size was insufficient to assess the more distal effects at 1-week follow-up.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes